CLINICAL TRIAL: NCT06376097
Title: Implementation of a Lung Cancer Screening Program in a Public Service, Using Low-dose Tomography and Metabolomics Evaluation
Brief Title: Lung Cancer Screening Program Using Low-dose Tomography and Metabolomic Evaluation in a Public Service.
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5162R00036
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
Keywords: Observational; Lung Cancer; Screening;
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Observational study that aims to evaluate the implementation of a lung cancer screening program in a smoker population included in a public heath service.

DETAILED DESCRIPTION:
Patients' clinical data (recruited from the outpatient clinics and wards of Hospital das Clínicas from the Faculty of Medicine of Botucatu) will be collected in a specific form, developed to this work, containing the following data: demographic characteristics (name, age, sex, race, profession, marital status, monthly income and education), main diagnosis and diseases associated, assessment of comorbidities using the Charlson Index, and Hospital Health Scale.

Anxiety and Depression (HAD Scale), use of maintenance medications, history of smoking (active or not, calculation of smoking load), body composition (mass index body- BMI calculation) and pulse oximetry measurement. All patients included will undergo low-dose radiation tomography and spirometry. All patients active smokers, who wish to stop smoking, will be referred to the outpatient clinic smoking cessation. Specific measurements will be applied if there is a diagnosis of COPD by spirometry (the BODE Index questionnaires, Dyspnea Index-Medical Modified Research Council, TC6) and patients will be referred to the outpatient clinic specific COPD for follow-up in the service. Subsequently, the anxiety and depression assessments. The tracking protocol will follow the recommendations of repeat the low-dose radiation chest tomography every year, if normal, until complete two years of follow-up. In this case, the patient will be discharged from the tracking. If the patient presents changes in the tomography, follow-up protocol according to the size of the lesions will be carried out. Morbidity and mortality assessment will be carried out in patients diagnosed with lung cancer.

ELIGIBILITY:
Inclusion Criteria:

Age between 45 and 74 years old; Smoker with a smoking history of at least 30 pack-years or former smoker who has quit smoking for less than 15 years; Never having participated in a lung cancer screening program ; Signing of the free and informed consent form.

Exclusion Criteria:

Patients with chronic diseases (cardiovascular, pulmonary, hepatic, renal or metabolic) at an advanced stage that limit life expectancy or make it impossible to perform a curative surgical procedure; Patients being treated for tuberculosis or other granulomatous diseases; Patients diagnosed with previous neoplasm(s) that could develop lung metastases; Pregnant women; Patients who, for some reason, are unable to undergo low-dose chest computed tomography; Patients previously submitted to thoracic radiotherapy.

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the outpatient clinics and wards of the Hospital das Clínicas of the Faculty of Medicine of Botucatu (HCFMB). The estimated sample size is 1000 patients.
  All patients recruited for this work who are diagnosed with a tobacco-related disease will be referred for outpatient monitoring and treatment of their pathologies. In addition, active smokers who wish to do so will be offered the Smoking Cessation Program.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2026-06-29 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Absolute number and frequency of false-negative lung nodules . | Dec, 2024
  Determine the prevalence of pulmonary nodules identified in the target population and the rate of false negative ones. Patients with suspicious nodules will be referred for transthoracic biopsy guided by tomography or a surgical biopsy.

SECONDARY OUTCOMES:
Assess adherence to smoking cessation treatment in active smokers who enter screening. | Dec, 2024
  Adherence to smoking cessation treatment will be objectively measured by the following calculation: number of smokers who stopped smoking after inclusion in the screening project / total number of mokers included. Information on smoking cessation will be extracted from the patient's medical record, from medical appointment carried out by the pulmonology team.
Assessment of morbidity and mortality in patients undergoing invasive procedures, whether diagnostic or therapeutic. | Dec, 2024
  The evaluation of morbidity and mortality will be objectively measured by the following calculations:
  -Morbidity: number of individuals who underwent an invasive procedure and who had complications / number of individuals who underwent an invasive procedure.
  Mortality: number of individuals who underwent an invasive procedure and died due to the procedure or a later compliaction / number of individuals who underwent an invasive procedure.
  Examples of complications after such procedures are: pneumonia after bronchoscopy or surgical procedures, pneumothorax and bleeding after bronchoscopy, surgical wound infection after surgical procedures, pneumothorax and hemothorax after transthoracic biopsy and death resulting from any invasive procedure
Cost comparasion of treating patients in metastatic setting vs. treating early-stage lung cancer patients, including all costs from the screening program. | Dec, 2024
  The costs of the screening program will comprise the following: medical consultations and by the multidisciplinary team, spirometry and CT scans. And when necessary, hospitalizations and invasive exams for the etiological investigation of the changes found in CT scans, such as bronchoscopy, transthoracic biopsy or surgical procedure.
  All costs from the program and treatment of early-stage diagnosed patients will be compared with a patient seen and treated in advanced stages of lung cancer (historical data). All costs will be estimated using data from hospital records.

CONTACTS AND LOCATIONS:
Overall Officials: Erica N Hasimoto, Principal Investigator — Hospital das Clínicas da Faculdade de Medicina de Botucatu (HCFMB)
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Botucatu (HCFMB), Botucatu, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/